CLINICAL TRIAL: NCT00769548
Title: A PHASE III TRIAL COMPARING WHOLE PELVIC IRRADIATION FOLLOWED BY A CONEDOWN BOOST TO BOOST IRRADIATION ONLY AND COMPARING NEOADJUVANT TO ADJUVANT TOTAL ANDROGEN SUPPRESSION (TAS)
Brief Title: Radiation Therapy and Hormone Therapy in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-9413; CDR0000063822
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-12

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Flutamide; Goserelin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 1 (Experimental): Neoadjuvant total androgen suppression (TAS) given 2 months before and during radiation therapy (RT) to the whole pelvis followed by a prostate boost.
  Interventions: Drug: flutamide; Drug: goserelin acetate; Radiation: low-LET photon therapy
- Arm 2 (Experimental): Neoadjuvant TAS given 2 months before and during RT to the prostate only.
  Interventions: Drug: flutamide; Drug: goserelin acetate; Radiation: low-LET photon therapy
- Arm 3 (Experimental): RT to the whole pelvis followed by a boost to the prostate followed by 4 months of TAS.
  Interventions: Drug: flutamide; Drug: goserelin acetate; Radiation: low-LET photon therapy
- Arm 4 (Experimental): RT to the prostate only followed by 4 months of TAS.
  Interventions: Drug: flutamide; Drug: goserelin acetate; Radiation: low-LET photon therapy

INTERVENTIONS:
Drug: flutamide — Drug used for TAS.
Drug: goserelin acetate — Drug used for TAS.
Radiation: low-LET photon therapy — radiation therapy
  Other Names: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high energy x-rays to damage tumor cells. Hormone therapy combined with radiation therapy may be a more effective treatment for prostate cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of four different combinations of radiation and hormone therapy in treating patients with prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Examine whether total androgen suppression (TAS) with flutamide/goserelin and whole-pelvic irradiation followed by a cone-down boost to the prostate improves progression-free survival at 5 years by at least 10% compared to TAS and prostate-only irradiation in patients with adenocarcinoma of the prostate at significant risk of nodal involvement. II. Examine whether induction and concurrent (neoadjuvant) TAS and radiotherapy improves the progression-free survival at 5 years by at least 10% compared to adjuvant TAS and radiotherapy. III. Compare treatments with regard to local control, time to distant failure, and overall survival.

OUTLINE: Randomized study. Arm I: Neoadjuvant Antiandrogen Therapy with Radiotherapy. Flutamide, FLUT, NSC-147834; Goserelin, Zoladex, ZDX, NSC-606864; with irradiation of the whole pelvis followed by a boost to the prostate using photons of at least 6 MV. Arm II: Neoadjuvant Antiandrogen Therapy with Radiotherapy; FLUT; ZDX; with irradiation of the prostate using equipment as in Arm I. Arm III: Radiotherapy followed by Adjuvant Antiandrogen Therapy. Irradiation as in Arm I; followed by FLUT; ZDX. Arm IV: Radiotherapy followed by Adjuvant Antiandrogen Therapy. Irradiation as in Arm II; followed by FLUT; ZDX.

PROJECTED ACCRUAL: 1,200 patients will be accrued over 2.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed adenocarcinoma of the prostate Any stage with an estimated risk of node involvement at least 15% (and therefore at significant risk for local and/or systemic failure) based on pretreatment PSA and Gleason score (GS), e.g.: GS of 7 and PSA greater than 7.5 ng/mL GS of 6 and PSA greater than 22.5 ng/mL GS of 5 and PSA greater than 37.5 ng/mL PSA greater than 4 and less than 100 ng/mL Highest pretreatment value determined by a monoclonal assay that has a normal range of 0-4 ng/mL PSA measured by polyclonal assay (e.g., Yang) that has a normal range of 0-2.5 ng/mL may need to be divided by a conversion factor of approximately 1.5 GS determination required prior to entry No distant metastases No biopsy proven lymph node involvement Ineligible for protocol RTOG-9408 (clinical stages T2c-T4 with GS of 6 or higher are eligible for this study)

PATIENT CHARACTERISTICS: Age: Any age Performance status: Karnofsky 70-100% Hematopoietic: Not specified Hepatic: Liver function tests no greater than 1.2 times normal Renal: Not specified Other: No major medical or psychiatric illness that would prevent completion of treatment or interfere with follow-up No second malignancy within 5 years except superficial nonmelanomatous skin cancer

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: At least 90 days since testosterone At least 60 days since finasteride Radiotherapy: No prior radiotherapy Surgery: No more than 60 days since surgical staging No radical surgery or cryosurgery

Max Age: 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1322 (Actual)
Dates: Start 1995-04; Primary Completion 2001-04 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (Arms 1, 3 vs. Arms 2, 4) | From randomization to the first occurrence of biochemical failure, clinical failure (local or distant), death from any cause, or last follow-up. Analysis occurs after all patients have been potentially followed for 5 years.

SECONDARY OUTCOMES:
Progression-free survival (Arms 1, 2 vs. Arms 3, 4) | From randomization to the first occurrence of biochemical failure, clinical failure (local or distant), death from any cause, or last follow-up. Analysis occurs after all patients have been potentially followed for 5 years.
Local progression | From randomization to the date of local progression or last follow-up. Analysis occurs after all patients have been potentially followed for 5 years.
Distant metastasis | From randomization to the date of metastatic disease or last follow-up. Analysis occurs after all patients have been potentially followed for 5 years.
Overall survival | From the date of randomization to the date of death or last follow-up. Analysis occurs after all patients have been potentially followed for 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Mack Roach, MD, Study Chair — University of California, San Francisco

REFERENCES:
- [Background] Du KL, Bae K, Movsas B, Yan Y, Bryan C, Bruner DW. Impact of marital status and race on outcomes of patients enrolled in Radiation Therapy Oncology Group prostate cancer trials. Support Care Cancer. 2012 Jun;20(6):1317-25. doi: 10.1007/s00520-011-1219-4. Epub 2011 Jul 1. PMID 21720747
- [Background] Hamstra DA, Bae K, Pilepich MV, Hanks GE, Grignon DJ, McGowan DG, Roach M, Lawton C, Lee RJ, Sandler H. Older age predicts decreased metastasis and prostate cancer-specific death for men treated with radiation therapy: meta-analysis of radiation therapy oncology group trials. Int J Radiat Oncol Biol Phys. 2011 Dec 1;81(5):1293-301. doi: 10.1016/j.ijrobp.2010.07.2004. Epub 2011 Mar 31. PMID 21458924
- [Background] Rodrigues G, Bae K, Roach M, Lawton C, Donnelly B, Grignon D, Hanks G, Porter A, Lepor H, Sandler H. Impact of ultrahigh baseline PSA levels on biochemical and clinical outcomes in two Radiation Therapy Oncology Group prostate clinical trials. Int J Radiat Oncol Biol Phys. 2011 Jun 1;80(2):445-52. doi: 10.1016/j.ijrobp.2010.02.034. Epub 2010 Aug 24. PMID 20615632
- [Background] Roach M 3rd, Bae K, Lawton C, Donnelly BJ, Grignon D, Hanks GE, Porter A, Lepor H, Venketesan V, Sandler H. Baseline serum testosterone in men treated with androgen deprivation therapy and radiotherapy for localized prostate cancer. Int J Radiat Oncol Biol Phys. 2010 Dec 1;78(5):1314-22. doi: 10.1016/j.ijrobp.2009.09.073. Epub 2010 Apr 8. PMID 20378270
- [Background] Millar J, Boyd R, Sutherland J. An update of the phase III trial comparing whole pelvic to prostate only radiotherapy and neoadjuvant to adjuvant total androgen suppression: updated analysis of RTOG 94-13, with emphasis on unexpected hormone/radiation interactions: in regard to Lawton et al. (Int J Radiat Oncol Biol Phys 2007;69:646-655.). Int J Radiat Oncol Biol Phys. 2008 May 1;71(1):316; author reply 316. doi: 10.1016/j.ijrobp.2008.01.009. No abstract available. PMID 18406900
- [Background] Williams S, Wiltshire K. Updated analysis of RTOG 94-13: in regard to Lawton et al. (Int J Radiat Oncol Biol Phys 2007;69:646-655). Int J Radiat Oncol Biol Phys. 2008 May 1;71(1):315; author reply 315-6. doi: 10.1016/j.ijrobp.2008.01.021. No abstract available. PMID 18406897
- [Background] Paner GP, Bae K, Grignon DJ, et al.: Trends in Gleason grading of prostate cancer (PCa): analysis of reporting by institutional and central review pathologists in four Radiation Therapy Oncology Group (RTOG) protocols spanning 17 years and 2094 needle biopsies (bxs). [Abstract] United States and Canadian Academy of Pathology 96th Annual Meeting, March 24-30, 2007, San Diego, CA. A-766, 2007.
- [Background] Pan CC, Bae K, Hanks GE, et al.: Comparison of two types of biochemical failures within the ASTRO and Phoenix Consensus definitions in patients treated on RTOG 92-02 and 94-13. [Abstract] Int J Radiat Oncol Biol Phys 66 (3 Suppl 1): A-2196, S318, 2006.
- [Background] Roach M, Moughan J, Movsas B, et al.: Socio-demographic predictors of biochemical failure and survival among high risk patients treated on Radiation Therapy Oncology Group (RTOG) prostate cancer trials: a meta-analysis. [Abstract] Int J Radiat Oncol Biol Phys 66 (3 Suppl 1): A-1127, S204, 2006.
- [Background] Ganswindt U, Paulsen F, Corvin S, Eichhorn K, Glocker S, Hundt I, Birkner M, Alber M, Anastasiadis A, Stenzl A, Bares R, Budach W, Bamberg M, Belka C. Intensity modulated radiotherapy for high risk prostate cancer based on sentinel node SPECT imaging for target volume definition. BMC Cancer. 2005 Jul 28;5:91. doi: 10.1186/1471-2407-5-91. PMID 16048656
- [Background] Johnke RM, Edwards JM, Evans MJ, Nangami GN, Bakken NT, Kilburn JM, Lee TK, Allison RR, Karlsson UL, Arastu HH. Circulating cytokine levels in prostate cancer patients undergoing radiation therapy: influence of neoadjuvant total androgen suppression. In Vivo. 2009 Sep-Oct;23(5):827-33. PMID 19779119
- [Background] Roach M 3rd. The role of PSA in the radiotherapy of prostate cancer. Oncology (Williston Park). 1996 Aug;10(8):1143-53; discussion 1154-61. PMID 8869957
- [Result] Lawton CA, DeSilvio M, Roach M 3rd, Uhl V, Kirsch R, Seider M, Rotman M, Jones C, Asbell S, Valicenti R, Hahn S, Thomas CR Jr. An update of the phase III trial comparing whole pelvic to prostate only radiotherapy and neoadjuvant to adjuvant total androgen suppression: updated analysis of RTOG 94-13, with emphasis on unexpected hormone/radiation interactions. Int J Radiat Oncol Biol Phys. 2007 Nov 1;69(3):646-55. doi: 10.1016/j.ijrobp.2007.04.003. Epub 2007 May 24. PMID 17531401
- [Result] Taussky D, Bae K, Bahary JP, Roach M 3rd, Lawton CA, Shipley WU, Sandler HM. Does timing of androgen deprivation influence radiation-induced toxicity? A secondary analysis of radiation therapy oncology group protocol 9413. Urology. 2008 Nov;72(5):1125-9. doi: 10.1016/j.urology.2007.11.067. Epub 2008 Mar 7. PMID 18314175
- [Result] Roach M 3rd, DeSilvio M, Valicenti R, Grignon D, Asbell SO, Lawton C, Thomas CR Jr, Shipley WU. Whole-pelvis, "mini-pelvis," or prostate-only external beam radiotherapy after neoadjuvant and concurrent hormonal therapy in patients treated in the Radiation Therapy Oncology Group 9413 trial. Int J Radiat Oncol Biol Phys. 2006 Nov 1;66(3):647-53. doi: 10.1016/j.ijrobp.2006.05.074. PMID 17011443
- [Result] Taussky D, Bae K, Bahary J, et al.: Does testosterone influence radiation-induced toxicity In radiotherapy of the prostate? A secondary analysis of RTOG protocol 9413. [Abstract] Int J Radiat Oncol Biol Phys 66 (3 Suppl 1): A-2215, S329-30.
- [Result] Roach M, DeSilvio M, Thomas C Jr, et al.: Field size and progression free survival (PFS) after neoadjuvant hormonal therapy (HT) and radiotherapy (RT) for prostate cancer: secondary analysis of RTOG 9413. [Abstract] American Society of Clinical Oncology 2005 Prostate Cancer Symposium, 17-19 February 2005, Orlando, Florida. A-87, 2005.
- [Result] Roach M, DeSilvio M, Thomas CR, et al.: Progression free survival (PFS) after whole-pelvic (WP) vs. mini-pelvic (MP) or prostate only (PO) radiotherapy (RT): a subset analysis of RTOG 9413, a phase III prospective randomized using neoadjuvant and concurrent (N&CHT). [Abstract] Int J Radiat Oncol Biol Phys 60 (Suppl 1): A-1014, S264, 2004.
- [Result] Roach M 3rd, DeSilvio M, Lawton C, Uhl V, Machtay M, Seider MJ, Rotman M, Jones C, Asbell SO, Valicenti RK, Han S, Thomas CR Jr, Shipley WS; Radiation Therapy Oncology Group 9413. Phase III trial comparing whole-pelvic versus prostate-only radiotherapy and neoadjuvant versus adjuvant combined androgen suppression: Radiation Therapy Oncology Group 9413. J Clin Oncol. 2003 May 15;21(10):1904-11. doi: 10.1200/JCO.2003.05.004. PMID 12743142
- [Result] Roach M III, DeSilvio M, Lawton C, et al.: Neoadjuvant hormonal therapy (NHT) with whole-pelvic (WP) radiotherapy (RT) improves progression-free survival (PFS): RTOG (Radiation Therapy Oncology Group) 9413, a phase III randomized trial. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-711, 2002.
- [Derived] Spratt DE, Tang S, Sun Y, Huang HC, Chen E, Mohamad O, Armstrong AJ, Tward JD, Nguyen PL, Lang JM, Zhang J, Mitani A, Simko JP, DeVries S, van der Wal D, Pinckaers H, Monson JM, Campbell HA, Wallace J, Ferguson MJ, Bahary JP, Schaeffer EM, Sandler HM, Tran PT, Rodgers JP, Esteva A, Yamashita R, Feng FY. Artificial Intelligence Predictive Model for Hormone Therapy Use in Prostate Cancer. NEJM Evid. 2023 Aug;2(8):EVIDoa2300023. doi: 10.1056/EVIDoa2300023. Epub 2023 Jun 29. PMID 38320143
- [Derived] Nguyen PL, Huang HR, Spratt DE, Davicioni E, Sandler HM, Shipley WU, Efstathiou JA, Simko JP, Pollack A, Dicker AP, Roach M, Rosenthal SA, Zeitzer KL, Mendez LC, Hartford AC, Hall WA, Desai AB, Rabinovitch RA, Peters CA, Rodgers JP, Tran P, Feng FY. Analysis of a Biopsy-Based Genomic Classifier in High-Risk Prostate Cancer: Meta-Analysis of the NRG Oncology/Radiation Therapy Oncology Group 9202, 9413, and 9902 Phase 3 Randomized Trials. Int J Radiat Oncol Biol Phys. 2023 Jul 1;116(3):521-529. doi: 10.1016/j.ijrobp.2022.12.035. Epub 2022 Dec 31. PMID 36596347
- [Derived] Spratt DE, Malone S, Roy S, Grimes S, Eapen L, Morgan SC, Malone J, Craig J, Dess RT, Jackson WC, Hartman HE, Kishan AU, Mehra R, Kaffenberger S, Morgan TM, Reichert ZR, Alumkal JJ, Michalski J, Lee WR, Pisansky TM, Feng FY, Shipley W, Sandler HM, Schipper MJ, Roach M 3rd, Sun Y, Lawton CAF. Prostate Radiotherapy With Adjuvant Androgen Deprivation Therapy (ADT) Improves Metastasis-Free Survival Compared to Neoadjuvant ADT: An Individual Patient Meta-Analysis. J Clin Oncol. 2021 Jan 10;39(2):136-144. doi: 10.1200/JCO.20.02438. Epub 2020 Dec 4. PMID 33275486
- [Derived] Roach M, Moughan J, Lawton CAF, Dicker AP, Zeitzer KL, Gore EM, Kwok Y, Seider MJ, Hsu IC, Hartford AC, Horwitz EM, Yamoah K, Jones CU, Michalski JM, Lee WR, Pisansky TM, Rabinovitch R, Rotman M, Pryzant RM, Kim HE, Thomas CR Jr, Shipley WU, Sandler HM. Sequence of hormonal therapy and radiotherapy field size in unfavourable, localised prostate cancer (NRG/RTOG 9413): long-term results of a randomised, phase 3 trial. Lancet Oncol. 2018 Nov;19(11):1504-1515. doi: 10.1016/S1470-2045(18)30528-X. Epub 2018 Oct 10. PMID 30316827